CLINICAL TRIAL: NCT00136903
Title: A Phase II, Randomized Study to Evaluate the Safety and Efficacy of Prochymal® (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) For the Treatment of Acute GVHD in Patients Who Receive Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Efficacy Study of Adult Human Mesenchymal Stem Cells to Treat Acute Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260-261; NCT00476762 (obsolete NCT alias)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Graft Vs Host Disease
Keywords: Graft vs Host Disease; (GVHD); Graft Versus Host Disease; Bone marrow transplant; Stem cells; Mesenchymal stem cells (MSCs); Adult stem cells; Leukemia; Lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma | interventions — remestemcel-l; Methylprednisolone; Prednisone; Cyclosporine; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochymal® - 2 Million cells/kg (Active Comparator): Participants will receive Prochymal® consisting of 2 million hMSCs/kg actual body weight, intravenously (IV) on Days 1 and 4 along with daily standard of care which includes methylprednisolone 2 milligrams (mg)/kg IV or prednisone 2.5 mg/kg orally. Participants will also continue cyclosporine, tacrolimus, and/or mycophenolate mofetil (MMF) at full therapeutic doses.
  Interventions: Drug: Prochymal® - 2 Million cells/kg; Drug: Methylprednisolone; Drug: Prednisone; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Prochymal® - 8 Million cells/kg (Active Comparator): Participants will receive Prochymal® consisting of 8 million hMSCs/kg actual body weight IV on Days 1 and 4 along with daily standard of care which includes methylprednisolone 2 mg/kg IV or prednisone 2.5 mg/kg orally. Participants will also continue cyclosporine, tacrolimus, and/or mycophenolate mofetil (MMF) at full therapeutic doses.
  Interventions: Drug: Prochymal®- 8 Million cells/kg; Drug: Methylprednisolone; Drug: Prednisone; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Prochymal® - 2 Million cells/kg — 2 million hMSCs/kg actual body weight, IV on study Days 1 and 4
  Other Names: Remestemcel-L; ex-vivo cultured adult human mesenchymal stem cells; hMSCs
  Arms: Prochymal® - 2 Million cells/kg
Drug: Prochymal®- 8 Million cells/kg — 8 million hMSCs/kg actual body weight IV on study Days 1 and 4
  Other Names: Remestemcel-L; ex-vivo cultured adult human mesenchymal stem cells; hMSCs
  Arms: Prochymal® - 8 Million cells/kg
Drug: Methylprednisolone — Methylprednisolone 2 mg/kg administered intravenously.
Drug: Prednisone — Prednisone 2.5 mg/kg administered orally.
Drug: Cyclosporine — Administered as prescribed by the caregiver.
Drug: Tacrolimus — Administered as prescribed by the caregiver.
Drug: Mycophenolate Mofetil — Administered as prescribed by the caregiver.

SUMMARY:
To establish the safety and efficacy of two dose levels of ex-vivo cultured adult human mesenchymal stem cells (hMSCs) (Prochymal®) in participants experiencing acute GVHD, Grades II-IV, post hematopoietic stem cells (HSC) transplant.

DETAILED DESCRIPTION:
Protocol 260 - Participants will be randomized with equal probability to the treatment arms (2 million cells/kilogram (kg) of Prochymal® or 8 million cells/kg of Prochymal®) using a stratified block design. The stratification factor is acute GVHD grade. For the purpose of stratification, the GVHD grades are II and III-IV. Treatment with investigational agent will be administered on study Days 1 and 4. Participants will be followed for safety and efficacy until Day 28 after initiation of treatment with the investigational agent, or until withdrawal or death, whichever occurs first.

Protocol 261- This study is designed as a long-term safety follow-up of participants who take part in the preceding clinical study of Prochymal® (Protocol 260) for the treatment of acute GVHD. Participants will be enrolled in Study 261 upon completion of the preceding Study 260.

ELIGIBILITY:
Protocol 260 Inclusion Criteria:

* Participant must be 18 to 70 years of age inclusive.
* If female and of child-bearing age, participant must be non-pregnant, not breast feeding, and use adequate contraception. Males must use adequate contraception.
* Participant must have newly diagnosed, Grade II-IV acute GVHD requiring therapy. Biopsy for confirmation of GVHD is not mandatory, but is recommended when feasible. Enrollment should not be delayed awaiting biopsy results.
* Participant must have received either full or reduced intensity myeloablative regimens followed by an allogeneic hematopoietic stem cell transplant using bone marrow, peripheral blood stem cell, or cord blood, including donor lymphocyte infusion (DLI).
* Participant must have minimal renal and hepatic function as defined by:

  * Calculated creatinine clearance (CLcr) of > 30 mL/min using the Cockroft-Gault equation.
* Participant must be available for all specified assessments at the study site through study Day 28.
* Participant must provide written informed consent and authorization for use and disclosure of protected health information (PHI).

Protocol 260 Exclusion Criteria:

* Participant has received previous treatment for Grade II-IV acute GVHD (except as noted in Criterion 2).
* Participant has been treated for GVHD with methylprednisolone, > 2mg/kg/day, for more than 72 hours prior to receiving Prochymal®.
* Participant has uncontrolled alcohol or substance abuse within 6 months of randomization.
* Participant has received an investigational agent (not approved by food and drug administration (FDA) for marketed use in any indication) within 30 days of randomization. Participant may not receive an investigational agent during the 28-day study period.
* Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant (e.g., uncontrolled infection, right heart failure, pulmonary hypertension, etc.).
* Participant has unstable arrhythmia.
* Participant is unwilling to sign consent form for the long-term follow-up study, Protocol 261.
* Participant has a known allergy to bovine or porcine products.
* Participant had received transplant for a solid tumor disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04-27 (Actual); Primary Completion 2006-07-28 (Actual); Study Completion 2008-07-14 (Actual)

PRIMARY OUTCOMES:
Protocol 260 - Response by Day 28, also called Overall Response (OR). OR includes complete response (CR) and partial response (PR) | 28 Days
Protocol 261-The incidence rate of different adverse events among participants treated with either dose of Prochymal® in the preceding study (Protocol No. 260). | 2 Years

SECONDARY OUTCOMES:
Protocol 260 - Partial Response or Improvement of GVHD by Day 28 in one or more organs involved with GVHD symptoms at Day 1, | 28 Days
Protocol 260 - Time to best response of GVHD | 28 Days
Protocol 260 - Time to improvement of GVHD in one or more organs | 28 Days
Protocol 261 - Survival through study day 90 | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, PA, Study Director — Mesoblast, Inc.
Locations (9):
- United States (9):
  - St. Francis Hospital, Indianapolis, Indiana
  - Kansas City Cancer Centers - BMT, Kansas City, Missouri
  - The Cancer Center at Hackensack University, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mt. Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - New York Medical College, Valhalla, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, FEC, Milwaukee, Wisconsin

REFERENCES:
- [Background] Bartholomew A, Sturgeon C, Siatskas M, Ferrer K, McIntosh K, Patil S, Hardy W, Devine S, Ucker D, Deans R, Moseley A, Hoffman R. Mesenchymal stem cells suppress lymphocyte proliferation in vitro and prolong skin graft survival in vivo. Exp Hematol. 2002 Jan;30(1):42-8. doi: 10.1016/s0301-472x(01)00769-x. PMID 11823036
- [Background] Deans RJ, Moseley AB. Mesenchymal stem cells: biology and potential clinical uses. Exp Hematol. 2000 Aug;28(8):875-84. doi: 10.1016/s0301-472x(00)00482-3. PMID 10989188
- [Background] Lazarus HM, Koc ON, Devine SM, Curtin P, Maziarz RT, Holland HK, Shpall EJ, McCarthy P, Atkinson K, Cooper BW, Gerson SL, Laughlin MJ, Loberiza FR Jr, Moseley AB, Bacigalupo A. Cotransplantation of HLA-identical sibling culture-expanded mesenchymal stem cells and hematopoietic stem cells in hematologic malignancy patients. Biol Blood Marrow Transplant. 2005 May;11(5):389-98. doi: 10.1016/j.bbmt.2005.02.001. PMID 15846293
- [Background] Le Blanc K, Rasmusson I, Sundberg B, Gotherstrom C, Hassan M, Uzunel M, Ringden O. Treatment of severe acute graft-versus-host disease with third party haploidentical mesenchymal stem cells. Lancet. 2004 May 1;363(9419):1439-41. doi: 10.1016/S0140-6736(04)16104-7. PMID 15121408
- [Background] Le Blanc K, Pittenger M. Mesenchymal stem cells: progress toward promise. Cytotherapy. 2005;7(1):36-45. doi: 10.1080/14653240510018118. PMID 16040382
- [Result] Kebriaei P, Isola L, Bahceci E, Holland K, Rowley S, McGuirk J, Devetten M, Jansen J, Herzig R, Schuster M, Monroy R, Uberti J. Adult human mesenchymal stem cells added to corticosteroid therapy for the treatment of acute graft-versus-host disease. Biol Blood Marrow Transplant. 2009 Jul;15(7):804-11. doi: 10.1016/j.bbmt.2008.03.012. PMID 19539211
- See also: Click here for more information on Prochymal® for treatment of GVHD — http://www.osiristx.com